CLINICAL TRIAL: NCT04297163
Title: Telemonitoring for the Recuperation of Patients With CPAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Jose M. Montserrat, Pneumologist consultor senior, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI17/01068
Record Dates: First submitted 2020-02-27; First posted 2020-03-05 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Telemedicine; Hospitals

STUDY DESIGN:
Intervention Model Description: 4-weeks randomized with parallel groups study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital management (Active Comparator): Patient's receive no intervention, the follow up is the usual for a patient following CPAP therapy.
  Interventions: Other: In Hospital
- Telemedicine management (Experimental): CPAP remote monitoring of patients, including a mobile application and a voicemail.
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — Remote CPAP monitoring, mobile app and voice mail
  Arms: Telemedicine management
Other: In Hospital — Face-to-face follow up
  Arms: Hospital management

SUMMARY:
This study is aimed at patients who do not achieve a minimum (≥4 hours/night) or optimal (≥5,5 hours/night) use of Continuous Positive Airway Pressure (CPAP) treatment and it is proposed to improve their adherence making a 4-weeks intervention using telemedicine tools: CPAP remote monitoring, a mobile application (app) and a voicemail. The concept of this work is to "recover" patients to minimum or optimal CPAP use.

DETAILED DESCRIPTION:
Given the prevalence of Obstructive Sleep Apnea (OSA), the symptoms it produces, which is a risk factor for various entities and that, in addition, its treatment clearly improves others; its control must be optimized in an effective and cost-effective manner. The use of information and communication technologies (ICT) in this context can be very beneficial.

The design of the study is prospective, randomized, controlled, open and parallel.

A ICT-based out of hospital management of OSA is implemented to be compared with the classical in-hospital management.

The main objectives were to evaluate the effectiveness of of two OSA management programs: the in-hospital classic management versus a telemedicine program based on the use of ICTs in the recovery of patients with OSA who who do not meet the minimum treatment (4 hours) or in those who do not comply with the optimal use (5.5 hours).

This is a 4-weeks management randomized, with parallel groups study. Participants will be patients from the Sleep Unit of Hospital Clinic Barcelona with OSA diagnosis and CPAP treatment indication, who after a follow-up between 3-months and up to 5 years have a CPAP compliance below 5,5 hours/night.

Two management programs will be compared:

* In-hospital classic management: Patients are followed regularly in the hospital with a face-to-face visit by the Sleep unit nurse.
* Telemedicine management: telemedicine support with mobile app, voicemail and CPAP remote monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* CPAP treatment initiated ≥1 month and <12 months
* CPAP compliance below 5.5 hours per night,
* Regular use of Smartphone and mobile apps.

Exclusion Criteria:

* Clinical suspicion or other confirmed sleep pathology,
* Severe nasal obstruction that prevents the use of CPAP,
* Physical-psychological inability to follow questionnaires and the program,
* Patients undergoing uvulopalatopharyngoplasty,
* Cheyne-Stokes syndrome,
* Pregnancy,
* Rejection in the initial test with CPAP during the training and education session and
* Failure to obtain informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
CPAP use | 4-weeks
  Compliance to CPAP treatment (Number of hours that the patient uses CPAP) will be taken as the main variable.

SECONDARY OUTCOMES:
Quality of life assessment | 4-weeks
  Functional Outcomes Sleep Questionnaire (FOSQ) and EuroQol-5D (EQ-5D)
Sleepiness assessment | 4 weeks
  Epworth sleepiness scale (ESS)
Satisfaction assessment | 4 weeks
  Satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Montserrat, Prof, Study Director — Hospital Clinic/Universitat de Barcelona
Locations (1):
- Josep M Montserrat Canal, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided